CLINICAL TRIAL: NCT00427323
Title: Disrupted Sleep in the Elderly: Light Exposure Studies
Brief Title: Light Exposure to Treat Sleep Disruption in Older People
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment has been put on hold until a future date
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG0076; 5R01AG006072-17 (NIH)
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2007-09

CONDITIONS: Sleep Initiation and Maintenance Disorders; Circadian Rhythm Sleep Disorders; Hypersomnia
Keywords: sleep; aging; biological rhythm; melatonin; alertness; early morning awakening; daytime sleepiness; difficulty maintaining sleep; sleep maintenance insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Disorders, Circadian Rhythm; Disorders of Excessive Somnolence

INTERVENTIONS:
Procedure: light exposure

SUMMARY:
The purpose of this study is to test whether shifts in the timing of the biological clock to a later hour (phase delay shifts of the human circadian system) can be produced in response to four successive evenings of light exposure, and whether that phase shift will result in greater evening alertness and greater nighttime sleep efficiency. Three different light sources will be compared: 1) standard fluorescent light; 2) blue-enriched light; 3) incandescent fluorescent light.

DETAILED DESCRIPTION:
The endogenous circadian pacemaker (the natural biological rhythm of a 24-hour cycle) is a major determinant of the timing of sleep and sleep structure in humans. There are considerable data from animals and humans suggesting that the properties of the circadian pacemaker change with advancing age. It has been hypothesized that these changes may underlie the sleep disruption and reduction in daytime alertness observed in the elderly. Recent studies have confirmed the impact of endogenous circadian phase on REM sleep (Rapid Eye Movement--the period of sleep associated with dreaming) and have revealed that high sleep efficiency can only be maintained when there is a unique phase-relationship between the sleep episode and endogenous circadian phase. This phase-relationship is such that even a small change in the relative timing of the circadian pacemaker and the daily sleep episode can have a large impact on an individual's ability to consolidate sleep throughout the night, especially in older individuals.

In this field-laboratory study, participants will first be monitored for 3 weeks while living at home on a self-selected sleep-wake schedule. They will then enter the laboratory for a 13-day study. The laboratory study begins with 3 baseline days living on their habitual schedule, and participants will be allowed to leave the hospital each day, returning in the evening. After this 3-day baseline, the initial circadian phase will be estimated in a constant posture (CP protocol). This is followed by a 4-day light treatment, when the participant will be exposed to approximately a 2 hour light session each evening. As in the baseline, the participant will be allowed to leave the hospital during the daytime hours, returning in the early evening. Following the 4-day treatment, a second CP will be conducted. After the CP, a 3-day laboratory follow up will take place (similar to the baseline), and this will be followed by an ambulatory follow-up, where the participant will be monitored with an actigraphy monitor for 3 weeks while living at home (as in the ambulatory baseline). Sleep will be polysomnographically recorded (oxygen saturation, electrocardiography, air flow, respiratory effort, limb movement, eye and jaw muscle movement, and brain electrical activity) each night in the laboratory, blood samples will be collected during each CP so that the phase of the circadian rhythm of melatonin secretion can be assessed, and activity monitoring will continue from the ambulatory baseline through the ambulatory follow-up. Tests of performance and alertness will be conducted during the times the participant is awake in the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Sleep complaint

Exclusion Criteria:

* Sleep apnea
* Depression
* Periodic limb movements of sleep
* Restless Legs Syndrome
* History of stroke
* History of heart attack
* Uncontrolled medical condition

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-06; Primary Completion 2007-09 (Estimated); Study Completion 2007-09 (Estimated)

PRIMARY OUTCOMES:
change in sleep efficiency
shift of circadian phase of melatonin secretion

SECONDARY OUTCOMES:
change in alertness and performance

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne F Duffy, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Duffy JF, Zeitzer JM, Czeisler CA. Decreased sensitivity to phase-delaying effects of moderate intensity light in older subjects. Neurobiol Aging. 2007 May;28(5):799-807. doi: 10.1016/j.neurobiolaging.2006.03.005. Epub 2006 Apr 18. PMID 16621166
- [Background] Duffy JF, Wright KP Jr. Entrainment of the human circadian system by light. J Biol Rhythms. 2005 Aug;20(4):326-38. doi: 10.1177/0748730405277983. PMID 16077152
- [Background] Klerman EB, Davis JB, Duffy JF, Dijk DJ, Kronauer RE. Older people awaken more frequently but fall back asleep at the same rate as younger people. Sleep. 2004 Jun 15;27(4):793-8. doi: 10.1093/sleep/27.4.793. PMID 15283016
- [Background] Duffy JF, Zeitzer JM, Rimmer DW, Klerman EB, Dijk DJ, Czeisler CA. Peak of circadian melatonin rhythm occurs later within the sleep of older subjects. Am J Physiol Endocrinol Metab. 2002 Feb;282(2):E297-303. doi: 10.1152/ajpendo.00268.2001. PMID 11788360
- [Background] Dijk DJ, Duffy JF, Czeisler CA. Age-related increase in awakenings: impaired consolidation of nonREM sleep at all circadian phases. Sleep. 2001 Aug 1;24(5):565-77. doi: 10.1093/sleep/24.5.565. PMID 11480654
- [Background] Klerman EB, Duffy JF, Dijk DJ, Czeisler CA. Circadian phase resetting in older people by ocular bright light exposure. J Investig Med. 2001 Jan;49(1):30-40. doi: 10.2310/6650.2001.34088. PMID 11217145
- [Background] Dijk DJ, Duffy JF, Czeisler CA. Contribution of circadian physiology and sleep homeostasis to age-related changes in human sleep. Chronobiol Int. 2000 May;17(3):285-311. doi: 10.1081/cbi-100101049. PMID 10841208
- [Background] Zeitzer JM, Daniels JE, Duffy JF, Klerman EB, Shanahan TL, Dijk DJ, Czeisler CA. Do plasma melatonin concentrations decline with age? Am J Med. 1999 Nov;107(5):432-6. doi: 10.1016/s0002-9343(99)00266-1. PMID 10569297
- [Background] Duffy JF, Dijk DJ, Klerman EB, Czeisler CA. Later endogenous circadian temperature nadir relative to an earlier wake time in older people. Am J Physiol. 1998 Nov;275(5 Pt 2):R1478-87. doi: 10.1152/ajpregu.1998.275.5.r1478. PMID 9791064
- [Background] Dijk DJ, Duffy JF, Riel E, Shanahan TL, Czeisler CA. Ageing and the circadian and homeostatic regulation of human sleep during forced desynchrony of rest, melatonin and temperature rhythms. J Physiol. 1999 Apr 15;516 ( Pt 2)(Pt 2):611-27. doi: 10.1111/j.1469-7793.1999.0611v.x. PMID 10087357
- [Background] Dijk DJ, Duffy JF. Circadian regulation of human sleep and age-related changes in its timing, consolidation and EEG characteristics. Ann Med. 1999 Apr;31(2):130-40. doi: 10.3109/07853899908998789. PMID 10344586